CLINICAL TRIAL: NCT04960189
Title: GB34 Acupuncture as Adjuvant in Early Phase of Medical Treatment of Mild Acute Cholecystitis
Brief Title: GB34 Acupuncture in Acute Cholecystitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nigde Omer Halisdemir University (Other)
Responsible Party: Principal Investigator, Alirıza Erdoğan, Principal Investigator, Nigde Omer Halisdemir University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 08.06.2021/32
Record Dates: First submitted 2021-07-06; First posted 2021-07-13 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2026-01

CONDITIONS: Acute Cholecystitis
MeSH Terms: conditions — Cholecystitis, Acute | interventions — Acupuncture Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Acupuncture (Experimental): GB34 acupuncture will be applied every day. Patients will receive standard medical treatment
  Interventions: Procedure: Acupuncture
- Controls (No Intervention): Patients will only receive standard medical treatment

INTERVENTIONS:
Procedure: Acupuncture — Acupuncture will be performed bilateral on fibular aspect of the leg, in the depression anterior and distal to the head of the fibula by using 0,25x50mm needles.
  Arms: Acupuncture

SUMMARY:
The purpose of this pilot study is to investigate the effects of GB34 acupuncture, performed as adjuvant to standard medical treatment, on clinical response and laboratory parameters of patients with a diagnosis of acute cholecystitis.

DETAILED DESCRIPTION:
Acute cholecystitis is a frequent complication of gallbladder stones. The prevalence of gallbladder stone is 10-15% and in 35% of patients complications and recurrent symptoms develop in their lifetime. Acute cholecystitis is one of the most frequently encountered acute surgical conditions. It is manifested in 3-10% of patients referred to emergency departments with complaints of abdominal pain.

Although the gold standard of therapy is laparoscopic cholecystectomy in symptomatic cholecystitis and related complications, more than 70% of patients respond well to medical treatment at first place. Actually, timing of cholecystectomy was studied extensively, yet is still debatable. Early cholecystectomy is the operation performed within 72 hours of the beginning of the symptoms. Delayed cholecystectomy is the operation performed 6 weeks after the suppression of the inflammation. Investigators perform early cholecystectomy is in cases with perforation and complication like gangrenous or emphysematous acute cholecystitis whereas delayed cholecystectomy is preferred in the remaining patients.

In fact it is known for some time that ear and body acupuncture have modulatory effects on motor functions of gallbladder and even provide some improvement in acute cholecystitis. Previously, studies demonstrating that GB34 has specific effects on the motility of bile ducts were published. More recently, researchers were able to demonstrate that GB34 electro acupuncture have positive effects on gall bladder wall thickness and on WBC levels, by using an experimental rabbit model of acute cholecystitis. Additional functional MR studies were used to distinguish the neural specificity of the acupuncture points. GB34 were found to induce a specific response pattern which is more significant in motor functions in brain. Furthermore it is known for decades that acupuncture other than point specific effects, triggers self-healing mechanisms of the body via endogen pathways.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed and hospitalised patients with mild acute cholecystitis

Exclusion Criteria:

* Pregnant women
* Immunosuppressive patients
* Patients with intermediate and severe acute cholecystitis
* Patients with acalculous acute cholecystitis
* Patients with uncontrolled diabetes mellitus
* Patients with collegen tissue diseases
* Patients with malignancies
* Patients who are using anti-coagulant or anti-aggregant medications
* Patients with blood diseases
* Patients with BMI>35

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2021-07-01 (Actual); Primary Completion 2025-12-10 (Actual); Study Completion 2025-12-10 (Actual)

PRIMARY OUTCOMES:
Perceived pain | From hospital admission (baseline) until hospital discharge, with VAS assessments performed every 12 hours, assessed up to a maximum of 168 hours.
  Measured by Visual Analog Scale scored between 0 and 10. Zero refers to no pain whereas 10 refers to the worst pain perceived by the patient.
Analgesic dosage | From hospital admission (baseline) until hospital discharge, assessed up to a maximum of 168 hours.
  Total dosage of analgesic administered in mg

SECONDARY OUTCOMES:
Guarding | At hospital admission (baseline) and every 24 hours until hospital discharge, assessed up to a maximum of 168 hours.
  presence or absence of abdominal guarding assessed by investigators. Guarding is defined as a spasm of muscles that minimizes the motion or agitation of sites that are affected by injury or disease.
Abdominal tenderness | At hospital admission (baseline) and every 24 hours until hospital discharge, assessed up to a maximum of 168 hours.
  presence or absence of abdominal tenderness assessed by investigators. Rebound tenderness refers to pain or discomfort after pressing on the patient's abdomen .
Oral intake | From hospital admission (baseline) until first tolerated oral intake, assessed up to hospital discharge (maximum 168 hours).
  if patients tolerate oral intake or not
Antibiotic dosage | From hospital admission (baseline) through hospital discharge, assessed up to a maximum of 168 hours
  Total antibiotic dose administered during hospitalization (mg)
Direct bilirubin | At hospital admission (baseline) and every 48 hours until hospital discharge, assessed up to a maximum of 168 hours
  Direct bilirubin levels expressed in mg/dL
Total bilirubin | At hospital admission (baseline) and every 48 hours until hospital discharge, assessed up to a maximum of 168 hours
  Total bilirubin levels expressed in mg/dL
Amylase | At hospital admission (baseline) and every 48 hours until hospital discharge, assessed up to a maximum of 168 hours
  Amylase levels expressed in U/L
GGT | At hospital admission (baseline) and every 48 hours until hospital discharge, assessed up to a maximum of 168 hours
  Gamma glutamyl transferase levels expressed in U/L
ALP | At hospital admission (baseline) and every 48 hours until hospital discharge, assessed up to a maximum of 168 hours
  Alkaline phosphatase levels expressed in U/L
ALT | At hospital admission (baseline) and every 48 hours until hospital discharge, assessed up to a maximum of 168 hours
  Alanine aminotransferase levels expressed in U/L
AST | At hospital admission (baseline) and every 48 hours until hospital discharge, assessed up to a maximum of 168 hours
  Aspartate aminotransferase levels expressed in IU/L
CRP | At hospital admission (baseline) and every 48 hours until hospital discharge, assessed up to a maximum of 168 hours
  C-reactive protein levels expressed in mg/L
PLT | At hospital admission (baseline) and every 48 hours until hospital discharge, assessed up to a maximum of 168 hours
  platelet count in microliter
LYM% | At hospital admission (baseline) and every 48 hours until hospital discharge, assessed up to a maximum of 168 hours
  percent of lymphocytes
NEU% | At hospital admission (baseline) and every 48 hours until hospital discharge, assessed up to a maximum of 168 hours
  percent of neutrophils
WBC | At hospital admission (baseline) and every 48 hours until hospital discharge, assessed up to a maximum of 168 hours
  White blood cell count in microliter
Hb | At hospital admission (baseline) and every 48 hours until hospital discharge, assessed up to a maximum of 168 hours
  Hemoglobin values expressed as g/dL

CONTACTS AND LOCATIONS:
Overall Officials: Alirıza Erdoğan, MD, Principal Investigator — Niğde Ömer Halisdemir University
Locations (1):
- Niğde Ömer Halisdemir University Training and Research Hospital, Niğde, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bouassida M, Zribi S, Krimi B, Laamiri G, Mroua B, Slama H, Mighri MM, M'saddak Azzouz M, Hamzaoui L, Touinsi H. C-reactive Protein Is the Best Biomarker to Predict Advanced Acute Cholecystitis and Conversion to Open Surgery. A Prospective Cohort Study of 556 Cases. J Gastrointest Surg. 2020 Dec;24(12):2766-2772. doi: 10.1007/s11605-019-04459-8. Epub 2019 Nov 25. PMID 31768828
- [Background] Arer IM, Yabanoglu H, Caliskan K. Can red cell distribution width be used as a predictor of acute cholecystitis? Turk J Surg. 2017 Jun 1;33(2):76-79. doi: 10.5152/turkjsurg.2017.3392. eCollection 2017. PMID 28740954
- [Background] Zhou ML, Jia WR, Wang JT, Wang P, Guo LH, Sui MH. [Effect of Electroacupuncture at "Yanglingquan" (GB 34) Acupoint on White Blood Cell Count and Gallbladder Wall Thickness in Rabbits with Acute Cholecystitis]. Zhen Ci Yan Jiu. 2015 Jun;40(3):233-7. Chinese. PMID 26237977
- [Background] Yeo S, Choe IH, van den Noort M, Bosch P, Jahng GH, Rosen B, Kim SH, Lim S. Acupuncture on GB34 activates the precentral gyrus and prefrontal cortex in Parkinson's disease. BMC Complement Altern Med. 2014 Sep 15;14:336. doi: 10.1186/1472-6882-14-336. PMID 25220656
- [Background] Na BJ, Jahng GH, Park SU, Jung WS, Moon SK, Park JM, Bae HS. An fMRI study of neuronal specificity of an acupoint: electroacupuncture stimulation of Yanglingquan (GB34) and its sham point. Neurosci Lett. 2009 Oct 16;464(1):1-5. doi: 10.1016/j.neulet.2009.08.009. Epub 2009 Aug 8. PMID 19666085
- [Background] Andersson S, Lundeberg T. Acupuncture--from empiricism to science: functional background to acupuncture effects in pain and disease. Med Hypotheses. 1995 Sep;45(3):271-81. doi: 10.1016/0306-9877(95)90117-5. PMID 8569551